CLINICAL TRIAL: NCT01517724
Title: Phase II Study of Bortezomib Consolidation After High Dose Therapy and Autologous Stem Cell Transplantation for Multiple Myeloma
Brief Title: Bortezomib Consolidation Trial
Acronym: BCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/08/0170
Record Dates: First submitted 2011-12-20; First posted 2012-01-25 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-03

CONDITIONS: Multiple Myeloma
Keywords: MM; HDT; ASCT; consolidation; bortezomib
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib consolidation (Experimental): Bortezomib administered once a week 1.3mg/sq m; maximum of 8 cycles (each cycle is 4 weeks)
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — 1.3mg/sq m, subcutaneous injection, days 1, 8, 15 and 22 of 28 day cycle; maximum of 8 cycles
  Other Names: Velcade

SUMMARY:
The aim of this trial is to determine whether bortezomib improves response and delays progression for multiple myeloma patients after high dose therapy and autologous stem cell transplant. It will also assess the effect of bortezomib treatment on patient bone health.

ELIGIBILITY:
Inclusion Criteria:

* MM patients who have received high dose Melphalan with ASCT 3-4 months prior to registration and have not progressed
* Age 18 - 70 years
* Life expectancy > 6 months
* Written informed consent
* Creatinine < 400µmol/L
* Bilirubin < 3x upper limit of normal
* WHO performance status 0-2
* Contraceptive precautions where appropriate

Exclusion Criteria:

* Received bortezomib previously
* On, or planned for, steroid therapy
* Poor performance status (ECOG ≥ 3)
* Disease progression at any stage
* Past history of polio, cord compression or other neurological condition resulting in persisting neurological deficit ≥ grade 2
* Severe hepatic impairment, indicated by bilirubin ≥ 3x upper limit of normal, or AST > 2.5x upper limit of normal
* Pregnant or lactating women
* Allergic reaction attributable to bortezomib or to compounds containing boron or mannitol
* Severe cardiovascular disease
* History of acute infiltrative pulmonary or pericardial disease
* History of hypotension or has decreased blood pressure
* Peripheral neuropathy ≥ grade 2, or neuropathic pain
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Received any drugs or agents that inhibit or induce CYP2C19 or CYP3A4 within 14 days before the first dose of bortezomib
* Need for therapy with concomitant CYP 3A4 or CYP2C19 inhibitors
* Have received an experimental drug or used an experimental medical device within 4 weeks before the planned start of treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-12; Primary Completion 2014-12 (Actual); Study Completion 2019-01-24 (Actual)

PRIMARY OUTCOMES:
Change in Disease response | At 6 and 12 months after ASCT consolidated by bortezomib therapy
  Disease response prior to consolidation with bortezomib will be compared with disease response at 6 and 12 months post ASCT.
Number of patients with adverse events | Up to 8 months after treatment start
  The number and percentage of patients who experience adverse events related to bortezomib treatment will be summarised for patients who received bortezomib consolidation after ASCT

SECONDARY OUTCOMES:
assess effect of bortezomib consolidation on bone health | At 1, 2, 3 and 9 months after start of treatment
  Summary of changes from baseline, after cycle 1,2 and 3 of bortezomib treatment and at the end of treatment for markers of bone formation and resorption
assess the effect of bortezomib consolidation on Minimal Residue Disease status | At 6 and 12 months post ASCT
determine progression free survival | At 2 years post ASCT
evaluate the quality of life for patients receiving bortezomib consolidation | Up to 8 months after treatment start

CONTACTS AND LOCATIONS:
Overall Officials: Kwee Yong, Principal Investigator — University College, London
Locations (1):
- University College London, London, United Kingdom